CLINICAL TRIAL: NCT04599543
Title: Clinical Trial for the Safety and Efficacy of IL3 CAR-T Cell Therapy for Patients With CD123 Positive Relapsed and/or Refractory Acute Myeloid Leukemia
Brief Title: IL3 CAR-T Cell Therapy for Patients With CD123 Positive Relapsed and/or Refractory Acute Myeloid Leukemia
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD123-001
Record Dates: First submitted 2020-10-21; First posted 2020-10-22 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; CAR T-cell therapy; CD123
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of IL3 CAR T-cells (Experimental)
  Interventions: Drug: IL3 CAR T-cells

INTERVENTIONS:
Drug: IL3 CAR T-cells — Each subject receive IL3 CAR T-cells by intravenous infusion
  Other Names: IL3 CAR-T cells injection

SUMMARY:
A Study of IL3 CAR-T Cell Therapy for Patients With CD123 Positive Relapsed and/or Refractory Acute Myeloid Leukemia.

DETAILED DESCRIPTION:
This is a single arm, open-label, single-center study. This study is indicated for relapsed or refractory CD123+ acute myeloid leukemia. The selections of dose levels and the number of subjects are based on clinical trials of similar foreign products. 36 patients will be enrolled. Primary objective is to explore the safety, main consideration is dose-related safety.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of CD123+ AML per the US National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines for Acute Myeloid Leukemia (2016.v1);
2. Relapsed or refractory CD123+ AML (meeting one of the following conditions):

   1. CR not achieved after standardized chemotherapy;
   2. CR achieved following the first induction, but CR duration is less than 12 months;
   3. Ineffectively after first or multiple remedial treatments;
   4. 2 or more relapses;
3. The number of primordial cells in bone marrow is > 5% (by morphology), and/or > 0.01% (by flowcytometry);
4. Total bilirubin ≤ 51 umol/L, ALT and AST ≤ 3 times of upper limit ofnormal, creatinine ≤ 176.8 umol/L;
5. Echocardiogram shows left ventricular ejection fraction (LVEF) ≥50%;
6. No active infection in the lungs, blood oxygen saturation in indoorair is ≥ 92%;
7. Estimated survival time ≥ 3 months;
8. ECOG performance status 0 to 2;
9. Patients or their legal guardians volunteer to participate in the studyand sign the informed consent.

Exclusion Criteria:

Subjects with any of the following exclusion criteria were not eligible for this trial:

1. History of craniocerebral trauma, conscious disturbance,epilepsy,cerebrovascular ischemia, and cerebrovascular, hemorrhagicdiseases;
2. Electrocardiogram shows prolonged QT interval, severe heart diseasessuch as severe arrhythmia in the past;
3. Pregnant (or lactating) women;
4. Patients with severe active infections (excluding simple urinarytractinfectionand bacterial pharyngitis);
5. Active infection of hepatitis B virus or hepatitis C virus;
6. Concurrent therapy with systemic steroids within 2 weeks prior toscreening, except for the patients recently or currently receiving in haledsteroids;
7. Previously treated with any CAR-T cell product or other genetically-modified T cell therapies;
8. Creatinine>2.5mg/dl, or ALT / AST > 3 times of normal amounts, or bilirubin>2.0 mg/dl;
9. Other uncontrolled diseases that were not suitable for this trial;
10. Patients with HIV infection;
11. Any situations that the investigator believes may increase the risk ofpatients or interfere with the results of study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-11-15 (Estimated); Primary Completion 2023-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after IL3 targeted CAR T-cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after IL3 targeted CAR T-cells infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Acute Myeloid Leukemia (AML), Overall response rate (ORR) | At Month 1, 3, 6, 12, 18 and 24
  Assessment of ORR (ORR = CR + CRi) at Month 6, 12, 18 and 24
AML, Overall survival (OS) | Up to 2 years after IL3 CAR-T cells infusion
  From the first infusion of IL3 CAR-T cells to death or the last visit
AML, Event-free survival (EFS) | Up to 2 years after IL3 CAR-T cells infusion
  From the first infusion of IL3 CAR-T cells to the occurrence of any event, including death, relapse or generelapse, disease progression (any one occurs first), and the last visit
Quality of life | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) scale [For item1-28: max score: 112, min score: 28, higher scores mean a better outcome; for item 28-29: max score: 14, min score: 2, higher scores mean a worse outcome] to measure Quality of life at Baseline, Month 1, 3, 6, 9 and 12
Activities of Daily Living (ADL) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using Activities of Daily Living (ADL) scale (Barthel Index) [max score: 100, min score: 0, higher scores mean a better outcome] at Baseline, Month 1, 3, 6, 9 and 12
Instrumental Activities of Daily Living (IADL) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment of Instrumental Activities of Daily Living (IADL) scale [max score: 56, min score: 14, higher scores mean a worse outcome] at Baseline, Month 1, 3, 6, 9 and 12
Hospital Anxiety and Depression Scale (HADS) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using Hospital Anxiety and Depression Scale (HADS) [max score: 42, min score: 0, higher scores mean a worse outcome] at Baseline, Month 1, 3, 6, 9 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital，College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No